CLINICAL TRIAL: NCT07017374
Title: Proteomic Analysis of Serum Samples After Cardiac Arrest: a TTM-trial Substudy
Status: Active, not recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/324
Record Dates: First submitted 2025-05-22; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Arrest (CA); Proteomics
Keywords: out-of-hospital cardiac arrest; heart arrest; proteomics; prognostication; hypothermic temperature control; targeted temperature management
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest | interventions — Hypothermia, Induced

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Proteomic analysis, targeted temperature management — Biobank serum samples from patients that were included in the TTM trial will be used for proteomic analysis. TTM trial randomised patients to targeted temperature management of 33 °C or 36 °C.

SUMMARY:
Cardiac arrest remains a large contributor to morbidity and mortality. Animal studies suggest an improvement in mortality and neurological function with hypothermia after cardiac arrest, a finding that could not be verified in large clinical trials such as Target Temperature Management after Out-of-hospital Cardiac arrest (TTM) trial. Multimodal neuroprognostication is an important tool for differentiating patients that will recover after cardiac arrest, and currently only one biomarker is in clinical use. The purpose of this study is to explore proteomics profiles in TTM trial patients in order to search for potential novel biomarkers, therapeutic targets, and to explore phenotypes of post-cardiac arrest syndrome.

DETAILED DESCRIPTION:
Background: A pilot study investigating proteomic profiles from 78 patients from the Target Temperature Management after Out-of-hospital Cardiac arrest (TTM) trial revealed 35 proteins associated to functional outcome, and six proteins associated to targeted temperature management at 33 °C. We plan to investigate proteomic profiles in the full cohort of the previously collected TTM-trial biobank. The aim is to stratify protein profiles based on survival, functional outcome, targeted temperature management, and MIRACLE2 score in order to search for potential novel biomarkers, therapeutic targets, and to explore phenotypes of post-cardiac arrest syndrome.

Methods: All patients with available serum samples at 24, 48, and/or 72 hours after return of spontaneous circulation will be included in the liquid chromatography and tandem mass spectrometry analysis using diaPASEF, combining data-independent-acquisition of spectra with parallel accumulation-serial fragmentation. Statistical analysis will include data normalisation, exploratory principal component analysis, and differential expression analysis. Changes in serum protein abundance will be analysed according to survival and binary functional outcome (modified Rankin Scale 0-3 vs. 4-6) at six-months after randomisation, randomisation to target temperature of 33 °C or 36 °C, and the MIRACLE2 score. Secondary stratifications will include sex, age, time to return of spontaneous circulation, shockable vs. non-shockable initial rhythm, circulatory shock on admission, and presumed cause of death.

Conclusion: This study will provide information about proteomic profiles after cardiac arrest and may give insight for identification of novel biomarkers for prediction of outcome.

ELIGIBILITY:
Inclusion Criteria as defined in the TTM trial (NCT01020916):

* Age ≥ 18 years old
* Out-of-hospital cardiac arrest (OHCA) of presumed cardiac cause
* Return of spontaneous circulation (ROSC)
* Unconsciousness (Glasgow Coma Score < 8) (patients not able to obey verbal commands) after sustained ROSC

Exclusion Criteria as defined in the TTM trial (NCT01020916):

* In-hospital cardiac arrest
* OHCA of presumed non-cardiac cause, e.g. after trauma or dissection/rupture of major artery OR Cardiac arrest caused by initial hypoxia (i.e. drowning, suffocation, hanging).
* Known bleeding diathesis (medically induced coagulopathy (e.g warfarin, clopidogrel) does not exclude the patient).
* Suspected or confirmed acute intracranial bleeding
* Suspected or confirmed acute stroke
* Unwitnessed asystole
* Known limitations in therapy and Do Not Resuscitate-order
* Known disease making 180 days survival unlikely
* Known pre-arrest CPC 3 or 4
* Temperature < 30°C on admission
* > 4 hours (240 minutes) from ROSC to screening
* Systolic blood pressure < 80 mm Hg in spite of fluid loading/vasopressor and/or inotropic medication/intra aortic balloon pump. If the systolic blood pressure (SBP) is recovering during the inclusion window (220 minutes) the patient can be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with an out-of-hospital cardiac arrest with presumed cardiac cause.
Sampling Method: Probability Sample
Enrollment: 682 (Actual)
Dates: Start 2025-05-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differential protein abundance | Differential protein abundance is evaluated 24, 48, and/or 72 hours after return of spontaneous circulation after cardiac arrest. Clinical outcomes are evaluated 180 days after cardiac arrest.
  Differential protein abundance will be acquired using proteomic analysis of serum samples. Protein abundance will be stratified in statistical analysis according to pre-specified clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Nielsen, Professor, MD, Principal Investigator — Lund University, Helsingborg hospital
Locations (1):
- Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The acquired mass spectrometry data, result files from peptide-centric analyses, spectral libraries, and other metadata will be deposited to the ProteomeXchange Consortium and made publicly available.
Time Frame: After publication
Access Criteria: Publicly available

REFERENCES:
- [Background] Nielsen N, Wetterslev J, al-Subaie N, Andersson B, Bro-Jeppesen J, Bishop G, Brunetti I, Cranshaw J, Cronberg T, Edqvist K, Erlinge D, Gasche Y, Glover G, Hassager C, Horn J, Hovdenes J, Johnsson J, Kjaergaard J, Kuiper M, Langorgen J, Macken L, Martinell L, Martner P, Pellis T, Pelosi P, Petersen P, Persson S, Rundgren M, Saxena M, Svensson R, Stammet P, Thoren A, Unden J, Walden A, Wallskog J, Wanscher M, Wise MP, Wyon N, Aneman A, Friberg H. Target Temperature Management after out-of-hospital cardiac arrest--a randomized, parallel-group, assessor-blinded clinical trial--rationale and design. Am Heart J. 2012 Apr;163(4):541-8. doi: 10.1016/j.ahj.2012.01.013. PMID 22520518
- [Background] Lileikyte G, Bakochi A, Ali A, Moseby-Knappe M, Cronberg T, Friberg H, Lilja G, Levin H, Arman F, Kjellstrom S, Dankiewicz J, Hassager C, Malmstrom J, Nielsen N. Serum proteome profiles in patients treated with targeted temperature management after out-of-hospital cardiac arrest. Intensive Care Med Exp. 2023 Jul 17;11(1):43. doi: 10.1186/s40635-023-00528-0. PMID 37455296
- [Background] Nielsen N, Wetterslev J, Cronberg T, Erlinge D, Gasche Y, Hassager C, Horn J, Hovdenes J, Kjaergaard J, Kuiper M, Pellis T, Stammet P, Wanscher M, Wise MP, Aneman A, Al-Subaie N, Boesgaard S, Bro-Jeppesen J, Brunetti I, Bugge JF, Hingston CD, Juffermans NP, Koopmans M, Kober L, Langorgen J, Lilja G, Moller JE, Rundgren M, Rylander C, Smid O, Werer C, Winkel P, Friberg H; TTM Trial Investigators. Targeted temperature management at 33 degrees C versus 36 degrees C after cardiac arrest. N Engl J Med. 2013 Dec 5;369(23):2197-206. doi: 10.1056/NEJMoa1310519. Epub 2013 Nov 17. PMID 24237006